CLINICAL TRIAL: NCT07328061
Title: Effect of Virtual Reality on Anxiety and Pain During Trans-vaginal Ultrasound for Endometriosis: A Prospective Randomized Controlled Study.
Brief Title: Virtual Reality for Anxiety and Pain Management in Transvaginal Ultrasound for Endometriosis
Acronym: VR Endo TVU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Zajicek, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0142-23-SMC
Record Dates: First submitted 2025-12-28; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Endometriosis
Keywords: Virtual reality; VR distraction; Transvaginal Ultrasound; TVUS; Anxiety; Pain
MeSH Terms: conditions — Endometriosis; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Participants Are randomized to undergo either transvaginal ultrasound with virtual reality distraction or standard transvaginal ultrasound without virtual reality. Each participant is assigned to a single study arm for the duration of the study.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR- TVUS Group (Experimental): Participants undergo TVUS while using immersive virtual reality distraction
  Interventions: Behavioral: Virtual reality - based distraction
- Contro Group - Standard TVUS (No Intervention): Participants undergo standard TVUS, without virtual reality or any additional distraction intervention.

INTERVENTIONS:
Behavioral: Virtual reality - based distraction — Participants use an immersive virtual reality headset during TVUS. The intervention consists of immersive three-dimensional (3D) VR distraction delivered a head-mounted display, allowing participants to engage with a computer-simulated virtual environment, with or without guided audio based mindfulness relaxation techniques. The intervention is designed to reduce pain and anxiety during US examination. Each session lasts approximately 10-15 minutes, and may include calming music or guided meditation audio
  Arms: VR- TVUS Group

SUMMARY:
The goal of this study to evaluate whether virtual reality (VR)-based technology, designed to promote relaxation and support pain self-management, can reduce anxiety and pain during trans-vaginal ultrasound (TVUS) for endometriosis.

Participants, women undergoing TVUS for endometriosis will be randomly assigned to either VR distraction group (VR-TVUS) or a standard examination group (control).

Anxiety and pain levels will be assessed immediately before and after the TVUS.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 50 years.
* Confirmed or suspected diagnosis of endometriosis.
* Scheduled to undergo transvaginal ultrasound examination.
* Ability to understand the study procedures and independently complete study questionnaires.
* Provided written informed consent.

Exclusion Criteria:

* History of epilepsy or seizure disorders.
* History of migraines.
* Visual or hearing impairment.
* Diagnosed anxiety disorders.
* Claustrophobia.
* Current symptoms of dizziness or nausea.
* Active respiratory tract infection.
* Any contraindication to transvaginal ultrasound examination.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level measured by State Anxiety Inventory (STAI-S)Anxiety levels are assessed using the Stating | From immediately before the TVUS to immediately after completion of the examination.
  Anxiety levels are assessed using the State Anxiety Inventory (STAI-S). It includes 20 items such as "I feel calm " and "I am tense ". Participates were instructed to circle the number that best describes how they felt at that moment from 1 to 4 (from "Not at all" to "Very much so"). The STAI-S questionnaire is scored by summing the responses to the individual items and the possible scores ranges from 20 to 80, where 20-37 refers to "no or low anxiety", 38-44 to "moderate anxiety", and 45-80 to "high anxiety" (45-80). The outcome measure is the change in STAI-S score from before to immediately after the TVUS examination

SECONDARY OUTCOMES:
Change in pain intensity measured by Visual Analog scale (VAS) | From immediately before the TVUS to immediately after completion of the examination.
  Pain intensity is assessed using a VAS . VAS is a self-reported measure of pain expressed as a number on a continuum between 1 ("no pain") and 10 ("worst pain").
Change in heart rate and blood pressure '(including mean arterial pressure) during TVUS | The outcome measure is the change in the heart rate and blood pressure from immediately before to immediately after the TVUS examination.
  Heart rate and blood pressure level are measured as objective measures of emotional distress and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Endometriosis Center, Sheba Medical Center, Ramat Gan, Central District, Israel

IPD SHARING:
Plan to Share IPD: No